CLINICAL TRIAL: NCT06966778
Title: A Double Blind, Randomized, Placebo Controlled Study to Evaluate the Efficacy of Oxybutynin Chloride Extended-Release Tablets to Improve Early Continence Recovery After Robotic Prostatectomy
Brief Title: Oxybutynin ER to Promote Early Continence Recovery After Robotic Prostatectomy: A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Synmosa Biopharma Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202412012MIPD
Record Dates: First submitted 2025-05-04; First posted 2025-05-13 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Localized Prostate Cancer; Postoperative Urinary Incontinence
Keywords: Localized Prostate Cancer; Robot-Assisted Radical Prostatectomy (RARP); Early Continence Recovery; Postoperative Urinary Incontinence; Oxybutynin Chloride; Extended-Release Tablets; Double-Blind Randomized Study; Placebo-Controlled Trial
MeSH Terms: interventions — Tablets

STUDY DESIGN:
Intervention Model Description: In this parallel assignment interventional study model, participants are randomly assigned to one of two groups, with each group receiving a different intervention:
  Treatment Group: Participants will receive oxybutynin chloride extended-release tablets (10 mg/day) to assess the impact of the drug on early continence recovery following robot-assisted radical prostatectomy (RARP) for localized prostate cancer.
  Control Group: Participants will receive a placebo (identical in appearance to the active drug) to compare the effects of oxybutynin chloride with no active intervention.
  Both groups will undergo the same follow-up protocol, with assessments of continence recovery, adverse events, and other outcomes conducted at multiple time points (e.g., pre-surgery, 10 days post-Foley catheter removal, and at 1, 3, 6, 9, and 12 months post-surgery). This study design allows for a direct comparison between the treatment and control groups, helping to determine the effective
Who Masked: Participant, Care Provider, Investigator
Masking Description: In this study, study coordinators and data analysts are also masked to ensure that there is no bias in the data collection and analysis process. This further ensures that the evaluation of outcomes, such as the effectiveness of the treatment and the assessment of adverse events, is unbiased and objective.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxybutynin chloride extended-release tablets 5mg/tab, 2 tab, PO, qd. (Experimental): Description: Participants in this arm will receive oxybutynin chloride extended-release tablets (10 mg/day) to assess its effectiveness in improving early continence recovery after robot-assisted radical prostatectomy (RARP) for localized prostate cancer.
  Intervention: Drug: Oxybutynin chloride extended-release tablets (10 mg/day).
  Interventions: Drug: Oxybutynin chloride extended-release tablets 5mg/tab, 2 tab, PO, qd.
- Control (Placebo Comparator): Description: Participants in this arm will receive placebo tablets, identical in appearance to the active drug, to compare the effects of oxybutynin chloride with no active intervention.
  Intervention: Placebo: Placebo tablets (identical in appearance to the active drug).
  Interventions: Drug: Placebo (2 tab), PO, qd.

INTERVENTIONS:
Drug: Oxybutynin chloride extended-release tablets 5mg/tab, 2 tab, PO, qd. — The intervention being studied is oxybutynin chloride extended-release tablets (Oxbu), a muscarinic antagonist that is used to manage overactive bladder symptoms, including urinary incontinence. In this study, it is specifically evaluated for its potential to improve early continence recovery following robot-assisted radical prostatectomy (RARP) in patients with localized prostate cancer.
  This formulation is an extended-release version of oxybutynin, which allows for a slower, sustained release of the drug over time, ensuring more consistent therapeutic effects with reduced side effects compared to immediate-release formulations. The intervention involves a daily dose of 10 mg, administered as two 5 mg tablets, to assess its impact on postoperative continence recovery.
  The key distinction of this intervention is its focus on improving continence recovery after prostate cancer surgery, specifically through its targeted use in early post-surgical recovery, making it different from othe
  Other Names: Oxybutynin Extended-Release Tablets; Oxbu; oxybutynin chloride extended-release tablet
  Arms: Oxybutynin chloride extended-release tablets 5mg/tab, 2 tab, PO, qd.
Drug: Placebo (2 tab), PO, qd. — placebo, which is designed to look identical to the active drug but contains no therapeutic ingredient.
  Arms: Control

SUMMARY:
The goal of this double-blind, randomized, placebo-controlled study is to evaluate whether oxybutynin chloride extended-release tablets can improve early continence recovery after robot-assisted radical prostatectomy (RARP) in patients with localized prostate cancer.

The main questions it aims to answer are:

[Does oxybutynin chloride improve continence recovery after RARP compared to a placebo?] [What are the predictors of continence recovery?]

Researchers will compare the treatment group (oxybutynin chloride 10 mg/day) with the control group (placebo) to assess differences in continence outcomes.

Participants will:

[Take the assigned medication (oxybutynin chloride or placebo) daily for 1-3 months until continence recovery.] [Complete surveys (e.g., IPSS, IIEF, ICIQ) at several time points post-surgery, including before surgery, 10 days after Foley catheter removal, and up to 12 months.] [Record any adverse events or concomitant medication use.]

Safety and tolerability will be monitored, and statistical analyses will determine the efficacy and predictors of continence. The study adheres to ethical principles, local regulations, and GCP guidelines.

DETAILED DESCRIPTION:
Extended Description of the Protocol This study is a double-blind, randomized, placebo-controlled clinical trial designed to evaluate the efficacy of oxybutynin chloride extended-release tablets (Oxbu) in improving early continence recovery following robot-assisted radical prostatectomy (RARP) in patients with localized prostate cancer.

Study Design and Structure

The study involves 135 patients, with 120 expected to complete all study procedures. Participants will be randomly assigned to one of two groups:

Treatment group: Receives 10 mg/day of oxybutynin chloride extended-release tablets.

Control group: Receives a placebo (identical in appearance to active drug). The treatment period lasts from 1 to 3 months, or until participants achieve complete continence, defined as no need for urinary pads and less than one episode of incontinence per week.

Intervention and Administration Dosage: Two tablets (5 mg each) taken orally once daily for both treatment and control groups.

Concomitant medications:

Prohibited: α-receptor blockers, cholinergics, and anticholinergics, among others.

Permitted: Acetaminophen and antacids, provided they are documented and do not interfere with the study objectives.

Data Collection and Efficacy Evaluation

Participants' continence outcomes will be assessed through standardized tools, including:

International Prostate Symptom Score (IPSS) International Index of Erectile Function (IIEF) International Consultation on Incontinence Questionnaire (ICIQ) Measurements will occur at baseline (pre-surgery), 10 days post-Foley catheter removal, and at intervals up to 12 months post-surgery.

Safety Monitoring All adverse events (AEs) will be recorded, with severity and relationship to the study medication assessed. AEs will be documented in Case Report Forms (CRFs) and reviewed for safety monitoring.

Statistical Analysis

Statistical analysis will involve:

Continuous variables: Assessed using independent t-tests or Mann-Whitney U tests.

Categorical variables: Compared via chi-squared, Fisher's exact tests, or linear-by-linear association tests.

Predictor analysis: Logistic regression (univariate and multivariate). Significance: p-values < 0.05. Ethical Considerations The study complies with the Declaration of Helsinki, Good Clinical Practice (GCP), and local regulations. Ethical committee approval is required before enrolling participants, and all patients must provide written informed consent prior to participation.

Timeline Enrollment period: 12 months. Treatment duration: 1-3 months. Study completion: Approximately 42 months. This extended protocol description highlights key technical aspects, intervention methods, and analytical strategies while avoiding duplication of eligibility and outcome measures previously outlined.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Patients with localized prostate cancer who are scheduled to undergo robot-assisted radical prostatectomy (RARP).
* Age: Participants must be 18 years or older, with no upper age limit.
* Consent: Participants must provide written informed consent before undergoing any study procedures.
* Ability to Follow Protocol: Participants must be able to follow the protocol procedures throughout the study.

Exclusion Criteria:

* Surgical Complications: Participants who experience surgical complications during or after RARP requiring extraordinary medical or surgical treatment.
* Other Urinary Conditions: Participants with other diseases causing lower urinary tract symptoms (LUTS) or bladder pain, including:
* - Benign prostatic hyperplasia (BPH), chronic prostatitis, interstitial cystitis, painful bladder syndrome, or urinary tract infection.
* - Overactive bladder or any other condition affecting bladder function.
* Chronic Medication: Participants with long-term use of medications such as:
* - Alpha-blockers, antimuscarinics, or anticholinergics.
* Glaucoma: Participants with narrow-angle glaucoma.
* Urinary Retention: Participants with a history of urinary retention.
* Gastrointestinal Motility Issues: Participants with severe conditions affecting gastrointestinal motility.
* Concurrent Medications: Participants who are taking medications that are prohibited by the study protocol (e.g., cholinergic drugs, azole antifungals, smooth muscle relaxants).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2025-09-23 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Achieving Urinary Continence (0-1 Pad/Day) Within 12 Months After RARP | Up to 12 months post-surgery

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lim KT, Kim YT, Lee TY, Park SY. Effects of tamsulosin, solifenacin, and combination therapy for the treatment of ureteral stent related discomforts. Korean J Urol. 2011 Jul;52(7):485-8. doi: 10.4111/kju.2011.52.7.485. Epub 2011 Jul 24. PMID 21860770
- [Background] Ho CH, Chang TC, Lin HH, Liu SP, Huang KH, Yu HJ. Solifenacin and tolterodine are equally effective in the treatment of overactive bladder symptoms. J Formos Med Assoc. 2010 Oct;109(10):702-8. doi: 10.1016/S0929-6646(10)60114-3. PMID 20970066
- [Background] Vardy MD, Mitcheson HD, Samuels TA, Wegenke JD, Forero-Schwanhaeuser S, Marshall TS, He W. Effects of solifenacin on overactive bladder symptoms, symptom bother and other patient-reported outcomes: results from VIBRANT - a double-blind, placebo-controlled trial. Int J Clin Pract. 2009 Dec;63(12):1702-14. doi: 10.1111/j.1742-1241.2009.02209.x. PMID 19930331
- [Background] Yakoubi R, Lemdani M, Monga M, Villers A, Koenig P. Is there a role for alpha-blockers in ureteral stent related symptoms? A systematic review and meta-analysis. J Urol. 2011 Sep;186(3):928-34. doi: 10.1016/j.juro.2011.04.061. Epub 2011 Jul 24. PMID 21791359
- [Background] Beddingfield R, Pedro RN, Hinck B, Kreidberg C, Feia K, Monga M. Alfuzosin to relieve ureteral stent discomfort: a prospective, randomized, placebo controlled study. J Urol. 2009 Jan;181(1):170-6. doi: 10.1016/j.juro.2008.09.026. Epub 2008 Nov 14. PMID 19013590
- [Background] Damiano R, Autorino R, De Sio M, Giacobbe A, Palumbo IM, D'Armiento M. Effect of tamsulosin in preventing ureteral stent-related morbidity: a prospective study. J Endourol. 2008 Apr;22(4):651-6. doi: 10.1089/end.2007.0257. PMID 18338955
- [Background] Park SC, Jung SW, Lee JW, Rim JS. The effects of tolterodine extended release and alfuzosin for the treatment of double-j stent-related symptoms. J Endourol. 2009 Nov;23(11):1913-7. doi: 10.1089/end.2009.0173. PMID 19814699
- [Background] Walz J, Epstein JI, Ganzer R, Graefen M, Guazzoni G, Kaouk J, Menon M, Mottrie A, Myers RP, Patel V, Tewari A, Villers A, Artibani W. A Critical Analysis of the Current Knowledge of Surgical Anatomy of the Prostate Related to Optimisation of Cancer Control and Preservation of Continence and Erection in Candidates for Radical Prostatectomy: An Update. Eur Urol. 2016 Aug;70(2):301-11. doi: 10.1016/j.eururo.2016.01.026. Epub 2016 Feb 2. PMID 26850969
- [Background] Heesakkers J, Farag F, Bauer RM, Sandhu J, De Ridder D, Stenzl A. Pathophysiology and Contributing Factors in Postprostatectomy Incontinence: A Review. Eur Urol. 2017 Jun;71(6):936-944. doi: 10.1016/j.eururo.2016.09.031. Epub 2016 Oct 6. PMID 27720536
- [Background] Salomon L. Re: Bianco FJ, Scardino PT, and Eastham JA: Radical prostatectomy: long-term cancer control and recovery of sexual and urinary function ("Trifecta") (Urology 66(5 suppl): 83-94, 2005). Urology. 2008 Feb;71(2):362. doi: 10.1016/j.urology.2005.12.053. No abstract available. PMID 18308133
- [Background] Ficarra V, Novara G, Rosen RC, Artibani W, Carroll PR, Costello A, Menon M, Montorsi F, Patel VR, Stolzenburg JU, Van der Poel H, Wilson TG, Zattoni F, Mottrie A. Systematic review and meta-analysis of studies reporting urinary continence recovery after robot-assisted radical prostatectomy. Eur Urol. 2012 Sep;62(3):405-17. doi: 10.1016/j.eururo.2012.05.045. Epub 2012 Jun 1. PMID 22749852
- [Background] Stanford JL, Feng Z, Hamilton AS, Gilliland FD, Stephenson RA, Eley JW, Albertsen PC, Harlan LC, Potosky AL. Urinary and sexual function after radical prostatectomy for clinically localized prostate cancer: the Prostate Cancer Outcomes Study. JAMA. 2000 Jan 19;283(3):354-60. doi: 10.1001/jama.283.3.354. PMID 10647798
- [Background] Donovan JL, Hamdy FC, Lane JA, Mason M, Metcalfe C, Walsh E, Blazeby JM, Peters TJ, Holding P, Bonnington S, Lennon T, Bradshaw L, Cooper D, Herbert P, Howson J, Jones A, Lyons N, Salter E, Thompson P, Tidball S, Blaikie J, Gray C, Bollina P, Catto J, Doble A, Doherty A, Gillatt D, Kockelbergh R, Kynaston H, Paul A, Powell P, Prescott S, Rosario DJ, Rowe E, Davis M, Turner EL, Martin RM, Neal DE; ProtecT Study Group*. Patient-Reported Outcomes after Monitoring, Surgery, or Radiotherapy for Prostate Cancer. N Engl J Med. 2016 Oct 13;375(15):1425-1437. doi: 10.1056/NEJMoa1606221. Epub 2016 Sep 14. PMID 27626365
- [Background] Hamdy FC, Donovan JL, Lane JA, Mason M, Metcalfe C, Holding P, Davis M, Peters TJ, Turner EL, Martin RM, Oxley J, Robinson M, Staffurth J, Walsh E, Bollina P, Catto J, Doble A, Doherty A, Gillatt D, Kockelbergh R, Kynaston H, Paul A, Powell P, Prescott S, Rosario DJ, Rowe E, Neal DE; ProtecT Study Group. 10-Year Outcomes after Monitoring, Surgery, or Radiotherapy for Localized Prostate Cancer. N Engl J Med. 2016 Oct 13;375(15):1415-1424. doi: 10.1056/NEJMoa1606220. Epub 2016 Sep 14. PMID 27626136